CLINICAL TRIAL: NCT04776629
Title: A Multi-Center, Randomized, Double-Blind, Placebo-controlled Proof-of-Activity Study With Orticumab in Subjects With Moderate-to-Severe Psoriasis and Cardiometabolic Risk Factors
Brief Title: A Proof-of-Activity Study With Orticumab in Subjects With Psoriasis and Cardiometabolic Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abcentra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ort-2020-01
Record Dates: First submitted 2021-02-16; First posted 2021-03-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Psoriasis; Inflammation; Coronary Artery Disease; Cardiometabolic Syndrome
MeSH Terms: conditions — Psoriasis; Inflammation; Coronary Artery Disease; Metabolic Syndrome | interventions — MLDL1278A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Active Comparator): Dosage: Repeating intravenous dose. Administered by infusion over 30 minutes.
  Frequency and duration: once weekly x 4 weeks, then once monthly x 2 months.
  Interventions: Drug: Orticumab
- Placebo (Placebo Comparator): Dosage: Repeating intravenous dose. Administered by infusion over 30 minutes.
  Frequency and duration: once weekly x 4 weeks, then once monthly x 2 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orticumab — A human recombinant monoclonal antibody against a specific oxidized low-density lipoprotein (oxLDL) epitope
  Other Names: MLDL1278a; BI-204; Anti-oxLDL Antibody
  Arms: Active Treatment
Drug: Placebo — Placebo for orticumab, containing all components of formulation except the active ingredient
  Arms: Placebo

SUMMARY:
The primary purpose of this proof-of-activity, phase 2 trial is to evaluate the safety and activity of orticumab in subjects with moderate to severe psoriasis and cardiometabolic risk factors.

DETAILED DESCRIPTION:
This randomized, double-blind, study is designed to compare the effect of orticumab against placebo in subjects with moderate to severe psoriasis and cardiometabolic risk factors. A total of 75 subjects will be randomized in a double-blind fashion to receive intravenous (IV) infusions either of orticumab or placebo for up to 78 days.

Participants will be enrolled into one of the two groups: active treatment or placebo. Subjects will be randomized in a 2:1 ratio, orticumab to placebo and receive up to 11 weeks of treatment.

Planned treatments are weekly x 4 , then monthly x 2 . The Internal Safety Review Committee (ISRC) will review the blinded safety data after the first subject completes the first dose (Day 1), the first five subjects complete the first dose (Day 1), and the first ten subjects complete the first dose (Day 1). The IRSC will review all adverse reactions to all administered doses at these times.

ELIGIBILITY:
Inclusion criteria:

* Stable/chronic plaque psoriasis with PASI score of ≥ 12 AND involving ≥ 10% of the subject's BSA.- ≥ 30 years of age at time of consent.
* BMI ≥ 30 kg/m2
* LDL ≥ 100 mg/dL at Screening.
* All females must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test prior to dosing.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria are met:

* Past use of orticumab.
* Any of the nonplaque forms of psoriasis: erythrodermic, guttate, or pustular.
* Scalp, palmar or plantar psoriasis only, at Screening or Baseline.
* Have evidence of skin conditions (e.g., eczema) at the time of Screening or Baseline visit that would interfere with theevaluation of psoriasis.
* Newly discovered Type 2 diabetes mellitus (T2DM)
* Moderate or high-intensity statin use or new use of a low-intensity statin therapy.
* No use of anti-coagulating or anti-thrombotic agents.
* Poorly controlled hypertension
* Use of an IL-23 blocker in the past 180 days, an IL-17 blocker in the past 16 weeks, or a TNF blocker in the past 12 weeks.
* Use of methotrexate, cyclosporine, or apremilast in the past 4 weeks.
* History of hypersensitivity or allergies to any contents in the orticumab formulation.
* A history of any clinically important abnormalities in cardiac rhythm or conduction.
* A history of prolonged QT intervals or a family history of long QT-syndrome at Screening.
* A history of first, second or third-degree atrioventricular (AV) block, or AV dissociation.
* A history of complete bundle branch block.
* Unstable angina pectoris, myocardial infarction, transient ischemic attack, or stroke within 3 months prior to Screening, or participants who have undergone percutaneous coronary intervention or a coronary artery bypass graft within 6 months prior to Screening or who are due to undergo these procedures at the time of Screening.
* Severe congestive heart failure (NYHA III or IV).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Mean percent change from Baseline in Psoriasis Area Severity Index (PASI) | 106 days (Week 15)
  PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
Percentage of participants achieving treatment success by the 5-point static Investigator's Global Assessment modified 2011 version (sIGA) Score | 106 days (Week 15)
  Percentage of participants achieving treatment success (clear =0 or almost clear =1) and greater than or equal to (>=) 2 Point Improvement at Week 15 on the sIGA scale
Incidence of Treatment Emergent Adverse Events (TEAEs) | 106 days (Week 15)
Incidence of serious adverse events (SAEs) | 106 days (Week 15)
Incidence of abnormal hemodynamic parameters | Weeks 3, 7, 11 and 15
  heart rate (HR) and blood pressure (BP)
Incidence of abnormal laboratory tests results | Weeks 3 and 15
Incidence of abnormal physical examination findings | Weeks 3, 7, 11, 15
  Physical examination will include the following organ or body system assessments: general appearance; eyes; ears, nose, and throat; head and neck; chest and lungs; cardiovascular; abdomen; musculoskeletal; lymphatic; dermatological; neurological; and extremities.

SECONDARY OUTCOMES:
Mean percent change from Baseline in Psoriasis Area Severity Index (PASI) | Weeks 1, 3, 7, and 11
  PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease)
Percentage of Participants achieving PASI75 and PASI50 | Weeks 1, 3, 7, and 11
  PASI75 is a 75 percent reduction in PASI score. PASI50 is a 50 percent reduction in PASI score
Mean percent change in Baseline in Body Surface Area (BSA) % involvement | Weeks 1, 3, 7, 11, 15
  Minimum: 0 percent, Maximum: 100 percent. Higher percentage indicates more skin with psoriasis.
Mean change from Baseline in Dermatology Life Quality Index (DLQI) score | Weeks 3, 7, 11, 15
  DLQI is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Mean change from Baseline in Itch Numerical Rating Scale (INRS) Score | Weeks 3 and 15
  The Itch NRS is a self-administered subject reported outcome questionnaire that is completed during protocol specified clinic visits. Participants indicate itch severity by circling the integer that best describes the worst level of itching due to psoriasis in the past 24 h on an 11-point scale anchored at 0, representing 'no itching' and 10, representing 'worst itch imaginable'.

OTHER OUTCOMES:
Change in Coronary Artery Inflammation by CCTA | 106 days (Week 15)
  Change in coronary artery perivascular fat attenuation index (FAI) measured by coronary computed tomographic angiography (CCTA)
Change in coronary artery plaque burden by CCTA | 106 days (Week 15)
  Change in total, noncalcified and low attenuation coronary artery plaque volume

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (13):
- United States (13):
  - CCT- Research at the center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Derm Institute & Skin Care Ctr., Inc., Santa Monica, California
  - Orange County Research Center, Tustin, California
  - Blue Coast Research Center, Vista, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - SMS Clinical Research, Mesquite, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, LTD.LLP, Webster, Texas
  - CCT Research - Springville Dermatology, Springville, Utah

REFERENCES:
- [Derived] Farina CJ, Davidson MH, Shah PK, Stark C, Lu W, Shirodaria C, Wright T, Antoniades CA, Nilsson J, Mehta NN. Inhibition of oxidized low-density lipoprotein with orticumab inhibits coronary inflammation and reduces residual inflammatory risk in psoriasis: a pilot randomized, double-blind placebo-controlled trial. Cardiovasc Res. 2024 May 29;120(7):678-680. doi: 10.1093/cvr/cvae057. No abstract available. PMID 38523341